CLINICAL TRIAL: NCT05140070
Title: Development and Implementation of an Innovative Technology for the Production New Generation Fruit and Vegetable Products Enriched With Dietary Fibre Preparation From Potato Starch With Prebiotic Properties for Children and Youth
Brief Title: Fruit and Vegetable Products Enriched With Fibre From Potato Starch With Prebiotic Properties for Children and Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Memorial Health Institute, Poland (Other)
Collaborators: Jan Dlugosz University in Czestochowa (Other); Tymbark MWS Sp. with o.o. Sp. K., Poland (Unknown); Faculty of Biotechnology and Food Sciences, Lodz University of Technology, Poland (Unknown); Oncology Center-Institute of Maria Skłodowska - Curie, Poland (Unknown)
Responsible Party: Principal Investigator, Piotr Socha, professor, Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PreSTFibre4kids
Record Dates: First submitted 2021-08-23; First posted 2021-12-01 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Overweight and Obesity; Child Obesity; Hypertension; NAFLD
Keywords: child; prebiotics; obesity; overweight; treatment
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity; Hypertension; Non-alcoholic Fatty Liver Disease | interventions — Vegetables; Diet

STUDY DESIGN:
Intervention Model Description: randomize, double blind, intervention vs control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the same appearance of the mousse (with and without active substance)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mousse with prebiotic
  Interventions: Dietary Supplement: Vegetable and fruit mousse enriched with a fiber preparation from potato starch with prebiotic properties; Behavioral: Dietary and physical activity counselling
- Control (Active Comparator): Mousse without prebiotic
  Interventions: Dietary Supplement: Vegetable and fruit mousse; Behavioral: Dietary and physical activity counselling

INTERVENTIONS:
Dietary Supplement: Vegetable and fruit mousse enriched with a fiber preparation from potato starch with prebiotic properties — All children in the intervention group will consume on daily basis vegetable and fruit mousse enriched with a fiber preparation from potato starch with prebiotic properties for six months
  Arms: Intervention
Dietary Supplement: Vegetable and fruit mousse — All children in the control group will consume on daily basis vegetable and fruit mousse for six months
  Arms: Control
Behavioral: Dietary and physical activity counselling — All children in the study will obtain 4 dietary and physical activity advice during the course of the study

SUMMARY:
The main goal of the project is to test fruit and vegetable mousse, with the addition of a fiber preparation made of potato starch with prebiotic properties, on selected clinical, metabolic and immunological parameters in overweight and obese children.

The study will be performed in a group of 80 to 100 children aged 6 to 10 years (pre-pubertal age), using a double-blind procedure. Children will be randomly assigned into two groups, i.e. the intervention group (they will receive a vegetable and fruit mousse with the addition of potato starch fiber preparation with prebiotic properties) and the control group (they will receive an identical preparation in their diet, but without the addition of potato starch fiber preparation).

DETAILED DESCRIPTION:
Purpose and nature of the study:

The study financed by the National Center for Research and Development is aimed at examining the vegetable and fruit mousse with the addition of a potato starch fiber preparation with prebiotic properties, in terms of preventing overweight and obesity in children and limiting the occurrence of metabolic disorders secondary to obesity.

Description of the procedures Children participating in the study will consume a daily fruit and vegetable mousse with or without the addition (control group) of a fiber-based potato starch preparation with prebiotic properties. Random selection will decide whether child will consume vegetable and fruit mousse with the addition of a fiber-based potato starch preparation with prebiotic properties. The study will be double blinded: neither parent and child, nor the attending physician will know whether the consumed mousse contains a fiber preparation. This method of conducting the study (random selection to the study group and control group and the so-called study blind) aims to eliminate the attitude of both the study participant and the observer to the therapy, which could affect the final assessment.

Children will take the mousse every day for six months (6 months). In order to evaluate the effect of fruit and vegetable mousse with the addition of a fiber preparation made of potato starch with prebiotic properties, the following tests will be performed: measurements of height, weight and, based on this measurements body mass index (BMI) will be calculated, waist circumference and blood pressure, bioimpedance test to assess the content of adipose and muscle tissue in the body, ultrasound of the carotid vessels and the liver, the speed of the pulse wave using the oscillometric method, the elastographic examination with a fibroscan, the examination of the composition of the intestinal flora in a stool sample, and a venous blood sample (7-10 ml volume) will be taken to evaluate lipid, carbohydrate metabolism, liver function, adipose tissue function, antioxidant status, and immune response parameters. The mentioned tests will be performed three times during the observation, i.e. at the time of enrollment in the study, after 6 months of taking the fruit and vegetable mousse and 3 months after the end of the vegetable and fruit mousse. In connection with participation in the study, the Child and Parents will be provided with dietary and physical activity advice as well as psychologist's advice on the day of enrollment in the study and at 3-month intervals up to 9 months from the start of participation in the study. Additionally, 3 months after starting taking the fruit and vegetable mousse, anthropometric and blood pressure measurements will be performed. During the participation in the study possible side effects will be registered.

A questionnaire containing questions about the child's date of birth, questions about the child's general health and taking medications, about the socio-demographic situation of the family, and food frequency questions will be completed.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obesity according to World Health Organization (WHO) definition
* in 20 patients additionally to overweight or obesity also increase blood pressure
* in 20 patients additionally to overweight or obesity also liver steatosis
* willingness to participate

Exclusion Criteria:

* allergy to mousse components
* malabsorption syndrome
* organ failure
* food neophobia
* other diseases or health problems which may interfere with study procedures or safety.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
BMI z-score change | 6 to 9 months
  Change in age and sex standardized BMI z-scores

SECONDARY OUTCOMES:
Bioimpedance | 6 to 9 months
  Change in body composition on bioimpedance (fat-body-mass %)
Waist | 6 to 9 months
  Change in waist z-score (cm)
Gut microbiota | 6 to 9 months
  change in microbiome composition
Triglyceride | 6 to 9 months
  change in triglyceride-parameter of lipid metabolism (mg%)
Cholesterol | 6 to 9 months
  change in cholesterol-parameter of lipid metabolism (mg%)
Low-density lipoprotein (LDL) | 6 to 9 months
  change in Low-density lipoprotein (LDL)-parameter of lipid metabolism (mg%)
high-density lipoprotein (HDL) | 6 to 9 months
  change in high-density lipoprotein (HDL)-parameter of lipid metabolism (mg%)
very low-density lipoprotein (VLDL) | 6 to 9 months
  change in very low-density lipoprotein (VLDL)-parameter of lipid metabolism (mg%)
apolipoprotein | 6 to 9 months
  change in apolipoprotein-parameter of lipid metabolism (mg%)
uric acid | 6 to 9 months
  change in uric acid (mg%)
leptin | 6 to 9 months
  change in leptin (ng/mL)
adiponectin | 6 to 9 months
  change in adiponectin (ng/mL)
glucose, serum | 6 to 9 months
  change in glucose (mg%)
insulin, serum | 6 to 9 months
  change in insulin (mcIU/mL)
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 6 to 9 months
  change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), score, normal range<2,5
Glutathione (GSH) | 6 to 9 months
  change in Glutathione (GSH) (g Hgb/mcL)
glutathione peroxidase (GPx) | 6 to 9 months
  change in glutathione peroxidase (GPx) (mg/dL)
total antioxidant status (TAS) | 6 to 9 months
  change in total antioxidant status (TAS) (mcmol/L)
tumor necrosis factor α (TNF-alfa) | 6 months
  change in tumor necrosis factor α (TNF-alfa) (ng/mL)
interleukin 6 (IL-6) | 6 months
  change in interleukin 6 (IL-6) (ng/mL)
Monocyte Chemoattractant Protein-1 (MCP-1) | 6 months
  change in Monocyte Chemoattractant Protein-1 (MCP-1) (ng/mL)
Macrophage Inflammatory Protein-1 (MIP-1) alfa and beta | 6 months
  change in Macrophage Inflammatory Protein-1 (MIP-1) alfa and beta (ng/mL)
Regulated upon Activation, Normal T Cell Expressed and Presumably Secreted (RANTES) | 6 months
  change in Regulated upon Activation, Normal T Cell Expressed and Presumably Secreted (RANTES) (ng/mL)
lymphocyte T | 6 months
  change in lymphocyte T (%)

CONTACTS AND LOCATIONS:
Locations (1):
- The Childen's Memorial Health Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data
URL: http://czd.pl

REFERENCES:
- [Result] Barczynska R, Kapusniak J, Litwin M, Slizewska K, Szalecki M. Dextrins from Maize Starch as Substances Activating the Growth of Bacteroidetes and Actinobacteria Simultaneously Inhibiting the Growth of Firmicutes, Responsible for the Occurrence of Obesity. Plant Foods Hum Nutr. 2016 Jun;71(2):190-6. doi: 10.1007/s11130-016-0542-9. PMID 27155867
- [Result] Barczynska R, Bandurska K, Slizewska K, Litwin M, Szalecki M, Libudzisz Z, Kapusniak J. Intestinal Microbiota, Obesity and Prebiotics. Pol J Microbiol. 2015;64(2):93-100. PMID 26373167
- [Result] Barczynska R, Slizewska K, Litwin M, Szalecki M, Kapusniak J. Effects of dietary fiber preparations made from maize starch on the growth and activity of selected bacteria from the Firmicutes, Bacteroidetes, and Actinobacteria phyla in fecal samples from obese children. Acta Biochim Pol. 2016;63(2):261-6. doi: 10.18388/abp.2015_1068. Epub 2016 Feb 29. PMID 26929930
- [Result] Litwin M, Sladowska J, Antoniewicz J, Niemirska A, Wierzbicka A, Daszkowska J, Wawer ZT, Janas R, Grenda R. Metabolic abnormalities, insulin resistance, and metabolic syndrome in children with primary hypertension. Am J Hypertens. 2007 Aug;20(8):875-82. doi: 10.1016/j.amjhyper.2007.03.005. PMID 17679036
- [Result] Litwin M, Michalkiewicz J, Trojanek J, Niemirska A, Wierzbicka A, Szalecki M. Altered genes profile of renin-angiotensin system, immune system, and adipokines receptors in leukocytes of children with primary hypertension. Hypertension. 2013 Feb;61(2):431-6. doi: 10.1161/HYPERTENSIONAHA.111.00181. Epub 2012 Dec 24. PMID 23266543
- [Result] Pinket AS, Van Lippevelde W, De Bourdeaudhuij I, Deforche B, Cardon G, Androutsos O, Koletzko B, Moreno LA, Socha P, Iotova V, Manios Y, De Craemer M; ToyBox-Study Group. Effect and Process Evaluation of a Cluster Randomized Control Trial on Water Intake and Beverage Consumption in Preschoolers from Six European Countries: The ToyBox-Study. PLoS One. 2016 Apr 11;11(4):e0152928. doi: 10.1371/journal.pone.0152928. eCollection 2016. PMID 27064274
- [Result] Socha P, Grote V, Gruszfeld D, Janas R, Demmelmair H, Closa-Monasterolo R, Subias JE, Scaglioni S, Verduci E, Dain E, Langhendries JP, Perrin E, Koletzko B; European Childhood Obesity Trial Study Group. Milk protein intake, the metabolic-endocrine response, and growth in infancy: data from a randomized clinical trial. Am J Clin Nutr. 2011 Dec;94(6 Suppl):1776S-1784S. doi: 10.3945/ajcn.110.000596. Epub 2011 Aug 17. PMID 21849603